CLINICAL TRIAL: NCT03339596
Title: Erythropoietin as an add-on Treatment for Cognitive Side-effects of Electroconvulsive Therapy
Brief Title: Effects of Erythropoietin for Cognitive Side-effects of ECT
Acronym: EPO-T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin Balslev Jørgensen (Other)
Collaborators: The Augustinus Foundation, Denmark. (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor-Investigator, Martin Balslev Jørgensen, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Organization: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-16038506; RHP-2017-023 (Other: The Danish Data Protection Agency Capital Region of Denmark); 2016-002326-36 (EudraCT Number)
Record Dates: First submitted 2017-10-24; First posted 2017-11-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: ECT; Cognitive Impairment; Unipolar Depression; Bipolar Depression
Keywords: electroconvulsive therapy; depression; cognition; cognitive side-effects; erythropoietin; functional magnetic resonance imaging
MeSH Terms: conditions — Cognitive Dysfunction; Depressive Disorder; Bipolar Disorder; Depression | interventions — Erythropoietin; Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythropoietin (Experimental): 4 intravenous infusions of recombinant human erythropoietin (EPO)
  Interventions: Drug: Erythropoietin
- Saline (Placebo Comparator): 4 intravenous infusions of saline (1 ml NaCl)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Erythropoietin — 40.000 IU/ml Erythropoietin (Epoetin alpha; Eprex) diluted with 100 ml saline (0.9% NaCl) is administered 4 times as intravenous infusions over 15 minutes.
  Other Names: Eprex; EPO
  Arms: Erythropoietin
Drug: Saline — 1 ml NaCl is administered 4 times as intravenous infusions over 15 minutes
  Other Names: Placebo
  Arms: Saline

SUMMARY:
EPO-T aims to investigate (i) whether short-term add-on treatment with erythropoietin (EPO) can reduce cognitive side-effects of ECT and (ii) whether such effects are long-lasting. Further, structural and functional magnetic resonance imaging (MRI) will be used to explore the neural underpinnings of such beneficial effects of EPO. Finally, the trial examines whether potential protective effects of EPO on cognition are accompanied by changes in markers of oxidative stress, inflammation, and neuroplasticity.

It is hypothesized that EPO treatment will (i) counteract ECT-induced cognitive decline, accompanied by (ii) increased sub-regional hippocampal volume, (iii) greater memory-related hippocampal activation and reinforcement of dorsolateral prefrontal activity during memory encoding and working memory, and (iv) changes in peripheral markers of inflammation, oxidative stress and neuroplasticity. Furthermore, we hypothesize that add-on EPO-treatment will produce greater, more sustained mood improvement than ECT treatment alone.

DETAILED DESCRIPTION:
The trial will include patients with a diagnosis of major depression (MDD) unipolar disorder (UD) or bipolar disorder (BD) with a current moderate to severe depressive episode symptoms (a score of >17 on the Hamilton Depression Rating Scale 17-items (HRDS-17) scheduled for ECT treatment. Patients will be recruited from Psychiatric Centres in The Mental Health Services in the Capital Region of Denmark and will undergo an eligibility assessment prior to randomization to 4 intravenous infusions of either recombinant human EPO (40.000 IU/ml; Epoetin alpha; Eprex, Janssen-Cilag) or placebo (1 ml NaCl) diluted with 100 ml saline (0.9% NaCl).

Cognitive functions, mood symptoms, and blood- and urine markers of inflammation, oxidative stress, and neuroplasticity will be assessed 3 times during the trial. First time at baseline, second time 3 days after ECT session 8 (patients skip one ECT session day after 8 ECTs to minimise the confounding effects of acute side-effects of ECT due to anaesthesia etc.), and the third time at a 3 month follow-up after ECT completion. In addition, the neuronal substrates for potential effects of EPO on cognition are investigated with structural and functional MRI after 8 ECT sessions (after 3 weekly EPO or saline infusions).

Block randomization and power calculations have been conducted by the independent Pharma Consulting Group AB (www.pharmaconsultinggroup.com). Treatment groups are stratified for age (>40 or <40) and gender.

The difference in cognitive change between EPO and saline-treated groups from baseline to post-treatment in our previous trial was 0.5 SD. Based on these findings, the sample size of N=52 (n=26 per group) in the current trial will reach a >0.8 power to detect a clinically relevant difference in the primary outcome measure (the cognitive composite score) between the 2 groups at an alpha level of 5% (two-sided test). The study is also powered to investigate differences in functional magnetic resonance imaging (fMRI) blood-oxygen dependent level (BOLD) response in key neural networks based on previous fMRI studies from our group in which sample sizes of 30 age and gender matched participants (n=15 per group) had the power of >0.8 to show drug-related effects on task-related neural response at an alpha level of p<0.05. In the current trial, inclusion of 52 participants (n=26 per treatment group) therefore ensures sufficient statistical power to detect EPO-related effects on neural activity.

Behavioural, mood, and biomarker data will be analysed using Mixed Models Design and Intention to Treat (ITT) approaches. Resting state and task-related fMRI data will be pre-processed and analyzed using FMRIB Expert Analysis Tool (FEAT) and the 'randomize' algorithm integrated in FSL, FMRIB Software Library (www.fmrib.ox.ac.uk/fsl).

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of major depressive disorder/unipolar disorder or bipolar disorder (confirmed using the Mini International Neuropsychiatric Interview; M.I.N.I.) with current moderate to severe depressive episode symptoms
* Hamilton Depression Rating Scale 17-items score ≥17
* Fluent Danish skills

Exclusion Criteria:

* Treatment under involuntary measures
* Other neuropsychiatric conditions
* Alcohol or substance misuse disorder
* Recent suicide attempts
* Diabetes
* Kidney disease
* Renal failure
* Untreated/insufficiently treated arterial hypertension
* Heart diseases (previously diagnosed or abnormal ECG findings during screening)
* Previous or current epilepsy in patient or first degree family
* Malignancies or thromboses
* Known allergy or antibodies against erythropoietin
* Initial hematocrit > 50% (males) or > 48% (females)
* Initial thrombocyte numbers over normal (>400 billions/L)
* Initial reticulocyte numbers <1‰
* Contraindications against prophylactic thrombosis treatment
* Myeloproliferative disorder, polycythemia
* Pregnancy or breast feeding
* Use of contraceptive medication or other hormonal contraceptives
* Sexually active women in the fertile age, who do not or do not want to use double barrier anticontraceptive methods
* Previous or current history of thromboembolic events or thromboses in patient or first degree family (increased risk of thromboembolic events)
* Overweight (BMI>30) or body weight <45 or >95 kg.
* Previous electroconvulsive therapy (ECT) treatment within last 3 months
* Reluctance or inability to comply with the protocol requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Cognitive composite score | Change from baseline to week 4 (i.e., after the last EPO injection and 8th ECT session)
  A cognitive composite score based on an average of the Rey Auditory Verbal Learning Test (RAVLT), The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding, Verbal Fluency with the letter "D", Wechsler Adult Intelligence Scale (WAIS)-III Letter-Number Sequencing, Trail Making Test Part B, and Rapid Visual Information Processing (RVP) from the Cambridge Neuropsychological Test Automated Battery (CANTAB Cognition Ltd.).

SECONDARY OUTCOMES:
Autobiographical Memory Interview-Short Form (AMI-SF) | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing retrograde autobiographical memory
Rey Auditory Verbal Learning Test (RAVLT) | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing verbal learning and memory

OTHER OUTCOMES:
Rey Auditory Verbal Learning Test (RAVLT) | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing verbal learning and memory
The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing attention
Verbal Fluency with the letter "D" | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing executive functions
Wechsler Adult Intelligence Scale (WAIS)-III Letter-Number Sequencing | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing executive functions
Trail Making Test Part B | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing executive functions
Rapid Visual Information Processing (RVP) from the Cambridge Neuropsychological Test Automated Battery (CANTAB Cognition Ltd.) | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Neuropsychological test assessing sustained attention
Hamilton Depression Rating Scale 17-items Version | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Clinician-based interview assessing depression severity
Beck Depression Inventory 21-items | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Questionnaire assessing subjectively-rated depression severity
Cognitive Complaints in Bipolar Disorder Rating Assessment | Baseline, week 4 (i.e., after the last EPO injection and 8th ECT session), and 3 months after ECT treatment completion
  Questionnaire assessing subjectively-rated cognitive complaints

CONTACTS AND LOCATIONS:
Overall Officials: Martin B. Jørgensen, Prof., Principal Investigator — Psychiatric Centre Copenhagen, Rigshospitalet; Kamilla W. Miskowiak, Prof., Study Director — Psychiatric Centre Copenhagen, Rigshospitalet
Locations (1):
- Mental Health Services, Capital Region of Denmark, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Copenhagen O, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miskowiak KW, Petersen JZ, Macoveanu J, Ysbaek-Nielsen AT, Lindegaard IA, Cramer K, Mogensen MB, Hammershoj LG, Stougaard ME, Jorgensen JL, Schmidt LS, Vinberg M, Ehrenreich H, Hageman I, Videbech P, Gbyl K, Kellner CH, Kessing LV, Jorgensen MB. Effect of erythropoietin on cognitive side-effects of electroconvulsive therapy in depression: A randomized, double-blind, placebo-controlled trial. Eur Neuropsychopharmacol. 2024 Feb;79:38-48. doi: 10.1016/j.euroneuro.2023.12.004. Epub 2023 Dec 20. PMID 38128460
- [Derived] Schmidt LS, Petersen JZ, Vinberg M, Hageman I, Olsen NV, Kessing LV, Jorgensen MB, Miskowiak KW. Erythropoietin as an add-on treatment for cognitive side effects of electroconvulsive therapy: a study protocol for a randomized controlled trial. Trials. 2018 Apr 19;19(1):234. doi: 10.1186/s13063-018-2627-2. PMID 29673379